CLINICAL TRIAL: NCT01467726
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Study of Safety, Pharmacokinetics and Pharmacodynamics of Velusetrag in Healthy Elderly Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of Velusetrag in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0048
Record Dates: First submitted 2011-10-28; First posted 2011-11-09 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2014-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Elderly
MeSH Terms: conditions — Alzheimer Disease | interventions — TD-5108

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose regimen 1 (Experimental): Varied doses
  Interventions: Drug: Velusetrag
- Dose regimen 2 (Experimental): Varied doses
  Interventions: Drug: Velusetrag
- Placebo (Experimental): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Velusetrag — Capsules
  Arms: Dose regimen 1
Drug: Velusetrag — Capsules
  Arms: Dose regimen 2
Drug: Placebo — Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 1, Randomized, Placebo-Controlled, Double-Blind, Study of Safety, Pharmacokinetics and Pharmacodynamics of Velusetrag in Healthy Elderly Subjects.

ELIGIBILITY:
Inclusion Criteria:

• Is in reasonably good health as determined by the investigator based on a detailed medical history, full physical examination (PE), vital signs (VS) (including blood pressure and pulse rate measurement), 12-lead ECG, and clinical laboratory tests.

* Subjects with mild, chronic, stable disease (e.g., controlled hypertension, controlled hypercholesterolemia, non-insulin dependent diabetes, osteoarthritis) may be enrolled if well controlled and not anticipated to interfere with the objectives of the study.
* Mild deviations from normal limits in PE, VS, ECG parameters, lab tests are acceptable if associated with the stable condition or are age-related

Exclusion Criteria:

* Has a condition, which in the opinion of the investigator, would confound or interfere with evaluation of safety and tolerability or PK or PD of the investigational drug, or prevent compliance with the protocol

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of repeat dosing of velusetrag | 3 weeks
  Number of subjects who complete the treatment period and are not withdrawn due to adverse events (AEs) or clinically significant findings on vital signs or ECGs

SECONDARY OUTCOMES:
Profile of Plasma Pharmacokinetics (PK) of velusetrag and metabolite | Days 1, 7, 8, 14, 15, 21 at predose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose and 24 hours postdose (and 48 and 72 h post Day 21 dose)
  Cmax (maximum observed concentration), Tmax (time of maximum observed concentration), AUC (area under the concentration-time curve)
Profile of urine PK of velusetrag and metabolite | Days 1, 7, 8, 14, 15, 21 0-24h postdose and 24-72 h post Day 21 dose
  Ae (amount excreted in urine), fe (fraction excreted in urine), CLr (renal clearance)
Pharmacodynamic effects of velusetrag | 3 weeks
  weekly bowel movement frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Development, Miramar, Florida, United States